CLINICAL TRIAL: NCT06996340
Title: Effects of White Noise on Pain, Anxiety and Comfort During in Invitro Fertilization: a Randomized Controlled Trial
Brief Title: White Noise and In-vitro Fertilizasyon
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yasemin Sökmen (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Yasemin Sökmen, Asistant Professor, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.30.2.ODM.0.20.08/718-772
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: WHITE NOISE, INVITRO FERTILIZATION, PAIN, ANXIETY, COMFORT
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: White noise group: The woman who was taken to the gynecological table for invirto fertilization will be made to listen to white noise (rain and waterfall sound) with a Bluetooth headset at a range of 75-85 decibels during the procedure. Because, it covers all sound ranges that people can hear within the range of 75-85 decibels (Cho and Hwang, 2021; Lin et al, 2018).
  Control group: The woman who was taken to the gynecological table for invirto fertilization was left to routine during the procedure.
Who Masked: Participant
Masking Description: White noise group: The woman who was taken to the gynecological table for invirto fertilization will be made to listen to white noise (rain and waterfall sound) with a Bluetooth headset at a range of 75-85 decibels during the procedure. Because, it covers all sound ranges that people can hear within the range of 75-85 decibels (Cho and Hwang, 2021; Lin et al, 2018).
  Control group: The woman who was taken to the gynecological table for invirto fertilization was left to routine during the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- White noise group: (Experimental): The woman who was taken to the gynecological table for invirto fertilization will be made to listen to white noise (rain and waterfall sound) with a Bluetooth headset at a range of 75-85 decibels during the procedure. Because, it covers all sound ranges that people can hear within the range of 75-85 decibels (Cho and Hwang, 2021; Lin et al, 2018).
  Interventions: Other: White noise group
- Control group: (Other): The woman who was taken to the gynecological table for invirto fertilization was left to routine during the procedure.
  Interventions: Other: routine care

INTERVENTIONS:
Other: White noise group — The woman who was taken to the gynecological table for invirto fertilization will be made to listen to white noise (rain and waterfall sound) with a Bluetooth headset at a range of 75-85 decibels during the procedure. Because, it covers all sound ranges that people can hear within the range of 75-85 decibels (Cho and Hwang, 2021; Lin et al, 2018).
  Arms: White noise group:
Other: routine care — routine care
  Arms: Control group:

SUMMARY:
In vitro fertilization is the placement of embryos into the uterus with a catheter under ultrasound guidance after the fertilization of sperm and oocytes in a laboratory tube. In the literature, various nonpharmacological methods such as acupuncture, yoga, meditation, deep breathing exercises, massage, art therapy and mind/body therapy have been used to cope with stress, pain and anxiety in infertile women. However, no study has been found examining the effect of white noise during in vitro fertilization. The aim of this study is to determine the effect of white noise on pain, anxiety and comfort during in vitro fertilization. This research is a randomized controlled experimental study. The universe of the study will consist of women coming to the in vitro fertilization center at Ondokuz Mayıs University Health Application and Research Center. The sample size of the study was calculated using the G*Power 3.1. 9.2 program, taking into account the data of the study by Fleury et al (2021). The post-procedure stress mean and standard deviation values of the experimental and control groups of the relevant study were used to calculate the effect size as 0.75. The minimum number of individuals to be included in the sample of this study was calculated using G*Power 3.1. 9.2 as effect size: 0.75, α= 0.05, power: 0.95, and the sample size was determined as 94 women (experimental group: 47, control group: 47). The data of the study will be collected with the Introduction Form, Visual Analog Scale, Anxiety Rating Scale, and General Comfort Scale Short Form. The data of the study will be evaluated using the SPSS 24 deviation, median and minimum-maximum values will be given. Chi-square test, Student t test, ANOVA test for those with normal distribution, Mann-Whitney U and Kruskal Wallis tests for those who are not.

DETAILED DESCRIPTION:
Assisted reproductive techniques are interventions that involve the in vitro processing of human oocytes, sperm or embryos for reproductive purposes (Zegers-Hochschild et al., 2017). In these interventions, various procedures such as ovarian stimulation, oocyte collection and embryo placement in the uterus are performed (Zhang et al., 2022). The most advanced and frequently used method of these procedures is in vitro fertilization. In in vitro fertilization, after the fertilization of sperm and oocyte in a tube in a laboratory environment, the resulting embryos are placed in the uterus with a catheter under ultrasound guidance (Çavuşoğlu, 2017). It has been reported that approximately 8 million children have been born since the initiation of procedures such as in vitro fertilization in the world (Fauser, 2019). Infertility is an important crisis in the lives of couples as it affects individuals physically, psychologically, emotionally, sexually and socially (Assaysh-Öberg et al, 2023; Kırca and Pasinlioğlu, 2019; Oh et al, 2024; Öztürk et al, 2020; Rooney and Domar, 2018). Because painful invasive procedures and interventions for diagnosis, uncertainty about the cause of infertility, lack of information about the treatment process, high cost of treatment, negative outcomes and social pressure lead to psychological problems in infertile individuals (Martínez-Pampliega et al, 2019; Oh et al, 2024; Öztürk et al, 2020; Rooney and Domar, 2018). The most common psychological problems are stress, anxiety and depression, and women experience stress before, during and after treatment (Kim et al, 2020; Kirca and Pasinlioglu, 2019; Rooney and Domar, 2018). The stress experienced both reduces the effectiveness of infertility treatment and causes treatment discontinuation (Kirca and Pasinlioglu, 2019; Rooney and Domar, 2018). In a study conducted on infertile women in Romania, it was reported that 63% of infertile women experienced stress during assisted reproductive treatment (Margan et al, 2022). Again, in a study examining the effect of stress on assisted reproductive treatment outcomes in infertile women in Tunisia, it was stated that women were much more stressed on the day of embryo transfer, and that primary infertile women had significantly higher stress levels than secondary infertile women (Sallem et al, 2021). There is a bidirectional and complex relationship between infertility and stress (Boivin, 2019). In addition, invasive procedures performed during the infertility diagnosis and treatment process cause pain, while the thought of whether the treatment will be successful or not causes stress (Assaysh-Öberg et al., 2023; de Boer et al., 2020). Health professionals need to support infertile women in coping with stress in order to reduce their stress levels (Rooney and Domar, 2018). When the studies in the literature are examined, different non-pharmacological methods such as acupuncture, yoga, meditation, deep breathing exercises, massage, art therapy and mind/body therapy have been used in infertile women to cope with stress (Akimbekov and Razzaque, 2021; Sis Çelik and Kırca, 2018; Gönül and Arslan, 2019; Kırca and Pasinlioğlu, 2019; Meier et al., 2021; Rooney and Domar, 2018). However, no study has been found examining the effect of white noise during in vitro fertilization. White noise is a continuous monotonous sound such as wind, waterfall, ocean waves or rain in the environment, and is a sound obtained by mixing equal amounts of different frequency sounds in a laboratory environment and preparing them in a digital environment and calibrating all of its frequencies (Cho and Hwang, 2021; Lin et al, 2018). Therefore, it was decided to conduct this study. The aim of this study is to determine the effect of white noise on pain, anxiety and comfort during in vitro fertilization.

Research Hypothesis; H01: There is no difference in pain between the white noise and control groups. H02: There is no difference in anxiety between the white noise and control groups.

H03: There is no difference in comfort between the white noise and control groups.

MATERIAL AND METHODS

Research Method

This research is a randomized controlled experimental research.

Place and Time of the Research

The research will be conducted in the in vitro fertilization center of a public university hospital in Samsun, Turkey, between January 2025 and August 2025.

Research Universe and Sample The research universe will consist of women who come to the in vitro fertilization center at the Ondokuz Mayıs University Health Application and Research Center. The sample size of the research was calculated using the G*Power 3.1.9.2 program, taking into account the data from the Fleury et al (2021) study. The effect size was calculated as 0.75 using the post-procedure stress mean and standard deviation values of the experimental and control groups of the relevant study. The minimum number of individuals to be included in the sample of this study was calculated using G*Power 3.1.9.2, effect size: 0.75, α= 0.05, power: 0.95, and the sample size was determined as 94 women (experimental group: 47, control group: 47). The group in which the participants would be included was determined using the full randomization technique on the website https://www.randomlists.com/team-generator (Figure 1).

3.947 / 5.000 Inclusion Criteria for the Study

Women between the ages of 18-35, diagnosed with primary infertility, not diagnosed with a psychiatric disease, able to speak and understand Turkish, and at least primary school graduates will be included in the study.

Exclusion Criteria for the Study Women who have undergone oocyte pick-up in the last month, intrauterine insemination in the last month, embryo transfer in the last month, or any other pharmacological or non-pharmacological application that can reduce stress will be excluded from the study.

Data Collection Tools The data of the study will be collected with the Introduction Form, Visual Analog Scale, Anxiety Assessment Scale, and General Comfort Scale Short Form.

Introduction form: This form was developed by the researchers based on the literature (Aba et al, 2017; Kalhori et al, 2020; Fleury et al, 2021). The form contains 17 questions in total, 13 of which include the socio-demographic characteristics of women (age, education level, employment status, spouse's age, spouse's education status, spouse's employment status, family type, place of residence, monthly income perception, etc.) and 4 questions include physiological parameters (blood pressure, pulse rate, respiratory rate, and oxygen saturation). The socio-demographic characteristics of women will be filled out in a face-to-face interview before the in vitro fertilization procedure, and the physiological parameters will be checked by the researcher before and after the procedure. Visual Analog Scale: It is a subjective scale used to evaluate different symptoms such as pain, satisfaction, allergic symptoms, anorexia, and anxiety (Berghmans Marten et al, 2017; Klimek et al, 2017; Mauri et al, 2015; Tashjian et al, 2017). This scale has a 10 cm horizontal line, one end of which indicates that the individual is "very good" and the other end is "very bad", and is evaluated by individuals by marking on it. This scale is expressed as "0 = I have no pain at all" and "10 = I have unbearable pain". The woman will be told that there are two extreme points and that she should mark any place between these points that matches the intensity of satisfaction. The distance between the beginning of "I am not satisfied at all" and this point marked by the woman will be measured and recorded in centimeters.

Anxiety Assessment Scale: The validity and reliability of the scale in Turkish was performed by Malakcıoğlu (2022). The scale has three sub-dimensions: physiological tension, worry and feeling insecure. There are a total of 10 items in the scale and it is evaluated as never, rarely, sometimes, often and almost always. The overall Cronbach's A internal consistency coefficients of the scale were calculated as 0.845, 0.770 in the physiological tension sub-dimension, 0.822 in the worry sub-dimension, and 0.838 in the feeling of insecurity sub-dimension. Malakcıoğlu (2022). General Comfort Scale Short Form: It was developed by Kolcaba (1992) and the validity and reliability of the scale were made by Çıtlık Sarıtaş et al (2018) (Çıtlık Sarıtaş et al, 2018). The scale has three sub-dimensions: relief, relaxation, and superiority. The scale consists of a total of 28 items and in the evaluation of the scale consisting of positive and negative items, the negative items are reverse coded and added. The average value is calculated by dividing the total score obtained by the number of scale items. The scale is scored between 1-6 and 6 points indicates a high level of comfort. In addition, the Cronbach alpha reliability coefficient of the Turkish form of the scale was 0.82, and the Cronbach alpha reliability coefficients of the sub-dimensions of the scale were calculated as relief 0.81, relaxation 0.81 and superiority 0.76 (Çıtlık Sarıtaş et al, 2018).

Preliminary Application A preliminary application will be conducted with five women to determine the understandability and applicability of the questionnaire form and the white noise application. If problems are detected regarding the understandability and application of the forms as a result of the preliminary application, the form will be revised.

Application of the Study Women who come to the IVF center for invirto fertilization, meet the inclusion criteria, and volunteer to participate in the study will be informed about the study and their written consent will be obtained. Before the invirto fertilization procedure, women will be interviewed face to face and their socio-demographic characteristics, preliminary results of physiological parameters and preliminary results of the anxiety assessment scale will be recorded in the questionnaire form. After the invirto fertilization procedure, physiological parameters will be re-evaluated by the researcher and the Visual Analog Scale, Anxiety Assessment Scale and General Comfort Scale Short Form will be filled out by women's own reporting.

White noise group: The woman who is taken to the gynecological table for invirto fertilization will be listened to white noise (rain and waterfall sound) with a Bluetooth headset in the range of 75-85 decibels during the procedure. Because, the range of 75-85 decibels covers all sound ranges that people can hear (Cho and Hwang, 2021; Lin et al, 2018).

Control group: The woman who was taken to the gynecological table for invirto fertilization was left to the routine during the procedure.

Evaluation of Data The data of the study will be evaluated using the Statistical Package for the Social Sciences 23 program. Percentage, arithmetic mean, standard deviation, median and minimum-maximum values will be used for descriptive statistics. All data will first be evaluated with Kolmogorov-Smirnov for compliance with normal distribution. In the analysis of the data, if the data have a normal distribution, Student t test and ANOVA will be applied, if not normally distributed, Mann Whitney U test and Kruskal Wallis will be applied. In the statistical evaluation, the significance level of the data will be taken as p<.05.

Ethical Aspect of the Research This research will be conducted in accordance with the principles of the Helsinki Declaration.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18-35,
* Diagnosed with primary infertility,
* Not diagnosed with a psychiatric disease,
* Who can speak and understand Turkish,
* Who are at least primary school graduates will be included in the study

Exclusion Criteria:

* Women who have undergone oocyte pick-up within the last month,
* Who have undergone intrauterine insemination within the last month,
* Who have undergone embryo transfer within the last month,
* Who have undergone any other pharmacological or non-pharmacological application that may reduce stress will be excluded.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women between the ages of 18-35 will be included in the study.
Enrollment: 94 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-06-02 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Pain | 30 minutes before in vitro fertilization
  Pain will be assessed with the Visual Analog Scale before and after the procedure.
Anxiety | 30 minutes before in vitro fertilization
  Will be evaluated with the Anxiety Assessment Scale.
Comfort | 30 minutes before in vitro fertilization
  It will be evaluated with the General Comfort Scale Short Form.

SECONDARY OUTCOMES:
Pain | 30 minutes after in vitro fertilization
  Pain will be assessed with the Visual Analog Scale before and after the procedure.
Anxiety | 30 minutes after in vitro fertilization
  Will be evaluated with the Anxiety Assessment Scale.
Comfort | 30 minutes after in vitro fertilization
  It will be evaluated with the General Comfort Scale Short Form.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Sökmen, Asistant professor, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aba YA, Avci D, Guzel Y, Ozcelik SK, Gurtekin B. Effect of music therapy on the anxiety levels and pregnancy rate of women undergoing in vitro fertilization-embryo transfer: A randomized controlled trial. Appl Nurs Res. 2017 Aug;36:19-24. doi: 10.1016/j.apnr.2017.05.005. Epub 2017 May 22. PMID 28720234
- [Background] Meier M, Wirz L, Dickinson P, Pruessner JC. Laughter yoga reduces the cortisol response to acute stress in healthy individuals. Stress. 2021 Jan;24(1):44-52. doi: 10.1080/10253890.2020.1766018. Epub 2020 May 26. PMID 32393092
- [Result] Akimbekov NS, Razzaque MS. Laughter therapy: A humor-induced hormonal intervention to reduce stress and anxiety. Curr Res Physiol. 2021;4:135-138. doi: 10.1016/j.crphys.2021.04.002. Epub 2021 Apr 30. PMID 34642668
- [Result] Infertility Workup for the Women's Health Specialist: ACOG Committee Opinion, Number 781. Obstet Gynecol. 2019 Jun;133(6):e377-e384. doi: 10.1097/AOG.0000000000003271. PMID 31135764
- [Result] Assaysh-Oberg S, Borneskog C, Ternstrom E. Women's experience of infertility & treatment - A silent grief and failed care and support. Sex Reprod Healthc. 2023 Sep;37:100879. doi: 10.1016/j.srhc.2023.100879. Epub 2023 Jun 20. PMID 37356208
- [Result] Bayu D, Egata G, Kefale B, Jemere T. Determinants of Infertility among Married Women Attending Dessie Referral Hospital and Dr. Misganaw Gynecology and Obstetrics Clinic, Dessie, Ethiopia. Int J Reprod Med. 2020 Mar 27;2020:1540318. doi: 10.1155/2020/1540318. eCollection 2020. PMID 32280671
- [Result] Berghmans JM, Poley MJ, van der Ende J, Weber F, Van de Velde M, Adriaenssens P, Himpe D, Verhulst FC, Utens E. A Visual Analog Scale to assess anxiety in children during anesthesia induction (VAS-I): Results supporting its validity in a sample of day care surgery patients. Paediatr Anaesth. 2017 Sep;27(9):955-961. doi: 10.1111/pan.13206. Epub 2017 Jul 14. PMID 28707384
- [Result] Boivin J. How does stress, depression and anxiety affect patients undergoing treatment? Curr Opin Obstet Gynecol. 2019 Jun;31(3):195-199. doi: 10.1097/GCO.0000000000000539. PMID 30893136
- [Result] Centers for Disease Control and Prevention [CDC]. (2023). Infertility FAQs. Centers for Disease Control and Prevention. https://www.cdc.gov/reproductivehealth/infertility/index.htm#:~:text =Yes.,to%20term%20(impaired%20fecundity (Erişim tarihi: 15.03.2023)
- [Result] Cho, M., Hwang, S. (2021). The effect of white noise on sleep in hospitalized patients: A randomized controlled trial. Korean Journal of Adult Nursing, 33(1), 44-55.
- [Result] Çavuşoğlu, İ., 2017. Yardımcı Üreme Teknikleri. İnfertilite Hemşireliği El Kitabı, Demirci, N. ve Beji, N.K. (editörler). Nobel Tıp Kitabevi, İstanbul, 103-120.
- [Result] Çıtlık, S. C., Çevik, S., Özden, G. (2018). Genel Konfor Ölçeği Kısa Formunun Türkçe geçerlik ve güvenirlik çalışması. Diyabet, Obezite ve Hipertansiyonda Hemşirelik Forumu Dergisi, 10(2), 16-22.
- [Result] de Boer ML, Bondevik H, Solbraekke KN. Beyond pathology: women's lived experiences of melancholy and mourning in infertility treatment. Med Humanit. 2020 Sep;46(3):214-225. doi: 10.1136/medhum-2018-011586. Epub 2019 Jun 6. PMID 31171635
- [Result] Estes SJ, Huisingh CE, Chiuve SE, Petruski-Ivleva N, Missmer SA. Depression, Anxiety, and Self-Directed Violence in Women With Endometriosis: A Retrospective Matched-Cohort Study. Am J Epidemiol. 2021 May 4;190(5):843-852. doi: 10.1093/aje/kwaa249. PMID 33184648
- [Result] Fauser BC. Towards the global coverage of a unified registry of IVF outcomes. Reprod Biomed Online. 2019 Feb;38(2):133-137. doi: 10.1016/j.rbmo.2018.12.001. Epub 2018 Dec 14. No abstract available. PMID 30593441
- [Result] Fleury EAB, Approbato MS, Barbosa MA. Interactive Music Therapy on Stress Level Reduction in Women Submitted to IVF/ICSI. Prospective Randomized Study. JBRA Assist Reprod. 2021 Apr 27;25(2):209-214. doi: 10.5935/1518-0557.20200068. PMID 33904665
- [Result] Gönül, K., Arslan, H., 2019. İnfertilite tedavisi alan çiftlerin kullandıkları tamamlayıcı ve alternatif tıp uygulamaları. Cukurova Medical Journal, 44, 329-338.
- [Result] Hudepohl NS, Smith K. Infertility and Its Association with Depression, Anxiety, and Emotional Distress: A Current Review, Advances in Psychiatry and Behavioral Health. 2022, 2(1), 119-132. https://doi.org/10.1016/j.ypsc.2022.05.005.
- [Result] Kalhori F, Masoumi SZ, Shamsaei F, Mohammadi Y, Yavangi M. Effect of Mindfulness-Based Group Counseling on Depression in Infertile Women: Randomized Clinical Trial Study. Int J Fertil Steril. 2020 Apr;14(1):10-16. doi: 10.22074/ijfs.2020.5785. Epub 2020 Feb 25. PMID 32112629
- [Result] Khizroeva J, Nalli C, Bitsadze V, Lojacono A, Zatti S, Andreoli L, Tincani A, Shoenfeld Y, Makatsariya A. Infertility in women with systemic autoimmune diseases. Best Pract Res Clin Endocrinol Metab. 2019 Dec;33(6):101369. doi: 10.1016/j.beem.2019.101369. Epub 2019 Dec 2. PMID 31837981
- [Result] Kirca N, Pasinlioglu T. The effect of yoga on stress level in infertile women. Perspect Psychiatr Care. 2019 Apr;55(2):319-327. doi: 10.1111/ppc.12352. Epub 2019 Jan 18. PMID 30657179
- [Result] Kim M, Moon SH, Kim JE. Effects of psychological intervention for Korean infertile women under In Vitro Fertilization on infertility stress, depression, intimacy, sexual satisfaction and fatigue. Arch Psychiatr Nurs. 2020 Aug;34(4):211-217. doi: 10.1016/j.apnu.2020.05.001. Epub 2020 May 5. PMID 32828351
- [Result] Klimek L, Bergmann KC, Biedermann T, Bousquet J, Hellings P, Jung K, Merk H, Olze H, Schlenter W, Stock P, Ring J, Wagenmann M, Wehrmann W, Mosges R, Pfaar O. Visual analogue scales (VAS): Measuring instruments for the documentation of symptoms and therapy monitoring in cases of allergic rhinitis in everyday health care: Position Paper of the German Society of Allergology (AeDA) and the German Society of Allergy and Clinical Immunology (DGAKI), ENT Section, in collaboration with the working group on Clinical Immunology, Allergology and Environmental Medicine of the German Society of Otorhinolaryngology, Head and Neck Surgery (DGHNOKHC). Allergo J Int. 2017;26(1):16-24. doi: 10.1007/s40629-016-0006-7. Epub 2017 Jan 19. PMID 28217433
- [Result] Kolcaba KY. Holistic comfort: operationalizing the construct as a nurse-sensitive outcome. ANS Adv Nurs Sci. 1992 Sep;15(1):1-10. doi: 10.1097/00012272-199209000-00003. PMID 1519906
- [Result] Liang S, Chen Y, Wang Q, Chen H, Cui C, Xu X, Zhang Q, Zhang C. Prevalence and associated factors of infertility among 20-49 year old women in Henan Province, China. Reprod Health. 2021 Dec 20;18(1):254. doi: 10.1186/s12978-021-01298-2. PMID 34930324
- [Result] Lin LW, Weng SC, Wu HS, Tsai LJ, Lin YL, Yeh SH. The Effects of White Noise on Agitated Behaviors, Mental Status, and Activities of Daily Living in Older Adults With Dementia. J Nurs Res. 2018 Feb;26(1):2-9. doi: 10.1097/JNR.0000000000000211. PMID 29315202
- [Result] Malakcioglu C. Validity and Reliability of the Anxiety Assessment Scale: A New Three-dimensional Perspective. Medeni Med J. 2022 Jun 23;37(2):165-172. doi: 10.4274/MMJ.galenos.2022.75318. PMID 35735160
- [Result] Margan R, Margan MM, Fira-Mladinescu C, Putnoky S, Tuta-Sas I, Bagiu R, Popa ZL, Bernad E, Ciuca IM, Bratosin F, Miloicov-Bacean OC, Vlaicu B, Dobrescu A. Impact of Stress and Financials on Romanian Infertile Women Accessing Assisted Reproductive Treatment. Int J Environ Res Public Health. 2022 Mar 10;19(6):3256. doi: 10.3390/ijerph19063256. PMID 35328944
- [Result] Martinez-Pampliega A, Cormenzana S, Martin S, Navarro L. Marital functioning and treatment outcome in couples undergoing assisted reproduction. J Adv Nurs. 2019 Feb;75(2):338-347. doi: 10.1111/jan.13844. Epub 2018 Oct 7. PMID 30187521
- [Result] Mauri PA, Contini NN, Giliberti S, Barretta F, Consonni D, Negri M, Di Benedetto I. Intrapartum epidural analgesia and onset of lactation: a prospective study in an Italian birth centre. Matern Child Health J. 2015 Mar;19(3):511-8. doi: 10.1007/s10995-014-1532-x. PMID 24894732
- [Result] Nik Hazlina NH, Norhayati MN, Shaiful Bahari I, Nik Muhammad Arif NA. Worldwide prevalence, risk factors and psychological impact of infertility among women: a systematic review and meta-analysis. BMJ Open. 2022 Mar 30;12(3):e057132. doi: 10.1136/bmjopen-2021-057132. PMID 35354629
- [Result] Oh HR, Chung YJ, Do HJ. Group tele-art therapy intervention in women undergoing in vitro fertilization: A randomized control study. The Arts in Psychotherapy, 2024, 91, 102227. https://doi.org/10.1016/j.aip.2024.102227.
- [Result] Ozturk A, Aba YA, Sik BA. The relationship between stigma, perceived social support and depression in infertile Turkish women undergoing in vitro fertilization-embryo transfer. Arch Psychiatr Nurs. 2021 Oct;35(5):434-440. doi: 10.1016/j.apnu.2021.05.009. Epub 2021 Jun 15. PMID 34561056
- [Result] Rooney KL, Domar AD. The relationship between stress and infertility. Dialogues Clin Neurosci. 2018 Mar;20(1):41-47. doi: 10.31887/DCNS.2018.20.1/klrooney. PMID 29946210
- [Result] Saei Ghare Naz M, Ozgoli G, Sayehmiri K. Prevalence of Infertility In Iran: A Systematic Review And Meta-Analysis. Urol J. 2020 Jun 23;17(4):338-345. doi: 10.22037/uj.v0i0.5610. PMID 32281088
- [Result] Sallem A, Essoussi H, Mustapha HB, Zaouali M, Ajina M. Impact of psychological stress on the outcomes of assisted reproduction in Tunisian infertile women. Pan Afr Med J. 2021 Dec 21;40:250. doi: 10.11604/pamj.2021.40.250.32207. eCollection 2021. PMID 35233270
- [Result] Sis Çelik, A., Kırca, N., 2018. İnfertil kadınların uyguladıkları tamamlayıcı ve destekleyici bakım uygulamaları. Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi, 21, 178-188.
- [Result] Tashjian VC, Mosadeghi S, Howard AR, Lopez M, Dupuy T, Reid M, Martinez B, Ahmed S, Dailey F, Robbins K, Rosen B, Fuller G, Danovitch I, IsHak W, Spiegel B. Virtual Reality for Management of Pain in Hospitalized Patients: Results of a Controlled Trial. JMIR Ment Health. 2017 Mar 29;4(1):e9. doi: 10.2196/mental.7387. PMID 28356241
- [Result] Türkiye Nüfus ve Sağlık Araştırması (TNSA), 2018. https://hips.hacettepe.edu.tr/tr/2018_turkiye_nufus_ve_saglik_arastirmasi-55 (27.04.2022).
- [Result] Word Health Organization 2023. İnfertility. https://www.who.int/publications/i/item/978920068315 (30.04.2023).
- [Result] Zegers-Hochschild F, Adamson GD, Dyer S, Racowsky C, de Mouzon J, Sokol R, Rienzi L, Sunde A, Schmidt L, Cooke ID, Simpson JL, van der Poel S. The International Glossary on Infertility and Fertility Care, 2017. Hum Reprod. 2017 Sep 1;32(9):1786-1801. doi: 10.1093/humrep/dex234. PMID 29117321
- [Result] Zhang L, Shao H, Huo M, Chen J, Tao M, Liu Z. Prevalence and associated risk factors for anxiety and depression in infertile couples of ART treatment: a cross-sectional study. BMC Psychiatry. 2022 Sep 19;22(1):616. doi: 10.1186/s12888-022-04256-9. PMID 36123644